CLINICAL TRIAL: NCT06324006
Title: A Phase 1, Randomized, Double-blind, Parallel and Placebo-controlled Single and Multiple Ascending Dose Trial Investigating Safety, Tolerability and Pharmacokinetics of LIB-01 in Healthy Participants.
Brief Title: A Phase 1 Trial of LIB-01 in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dicot AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCT3934
Record Dates: First submitted 2023-09-20; First posted 2024-03-21 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a Phase I, double-blind, parallel-group, placebo-controlled, randomized first-in-human trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIB-01 (Experimental): LIB-01 oral suspension
  Interventions: Drug: LIB-01
- Placebo (Placebo Comparator): Placebo oral suspension
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LIB-01 — LIB-01 oral suspension
  Arms: LIB-01
Other: Placebo — Placebo oral suspension
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the safety, tolerability and pharmacokinetics of LIB-01 in healthy male participants. The main questions it aims to answer are:

* How safe and tolerable is LIB-01 when given once or repeatedly at different dose levels.
* What are the pharmacokinetic characteristics of LIB-01

Participants will receive LIB-01 and be followed up for safety and pharmacokinetics by:

* Adverse events
* ECG
* Blood sampling for laboratory parameters and pharmacokinetic analysis

ELIGIBILITY:
Inclusion Criteria

1. Provision of signed and dated written informed consent prior to any trial specific procedures.
2. Healthy male participant aged 18 to 65 years, inclusive.
3. Body mass index ≥ 18.5 and ≤ 30.0 kg/m2.
4. Medically healthy participant without abnormal clinically significant medical history, physical findings, vital signs, ECG and laboratory values.
5. Participants must be willing to use an acceptable form of contraception and refrain from donating sperm from the administration of IMP until 3 months after the administration of IMP. Any female partner of a non-vasectomised male participant who is of child-bearing potential must use an acceptable contraceptive method from at least 2 weeks prior to the administration of IMP to 4 weeks after the administration of IMP.
6. Understands the trial requirements.
7. MAD participants only: Mild to moderate erectile dysfunction.

Exclusion criteria

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the results or the participant's ability to participate in the trial.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the (first) administration of IMP.
3. Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the trial.
5. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to LIB-01.
6. History of priapism.
7. History of glaucoma.
8. History of Non-Arteritic Anterior Ischemic Optic Neuropathy.
9. History of prostatectomy or prostate surgery.
10. Bleeding deficiencies or ongoing anticoagulant therapy that would put the participant at risk.
11. Cardiac disease, including but not limited to uncontrolled hypertension; unstable angina; myocardial infarction or cerebrovascular accident.
12. Any positive result for serum hepatitis B surface antigen, hepatitis C antibodies and/or human immunodeficiency virus (HIV).
13. Abnormal vital signs.
14. Shortened QT interval corrected according to Fridericia (QTcF), prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant ECG abnormalities.
15. Use of oral, injectable, or topical pro-erectile drugs or supplements.
16. Use of nitrates.
17. Ongoing antiandrogen treatment.
18. Regular use of any prescribed or non-prescribed medications, within 2 weeks (Part I:SAD) or 4 weeks (Part II: MAD) prior to the (first) administration of IMP, except occasional intake of paracetamol, as well as nasal decongestants without cortisone, antihistamine or anticholinergics for a maximum of 10 days.
19. Planned treatment or treatment with another investigational drug.
20. Current smokers or users of nicotine products.
21. Positive screening result for drugs of abuse or alcohol.
22. History of alcohol abuse or excessive intake of alcohol.
23. Presence or history of drug abuse.
24. History of, or current use of anabolic steroids.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of treatment-emergent adverse events as assessed by CTCAE in healthy male participants, following a single oral dose of LIB-01. | 14 days
  Frequency, seriousness and intensity of adverse events. Adverse events will be graded from 1-5 by the Common Terminology Criteria for Adverse Events (CTCAE):
  Grade 1, Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2, Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL).
  Grade 3, Severe or medically significant but not immediately life-threatening; hospitalisation or prolongation of hospitalisation indicated; disabling; limiting self- care ADL.
  Grade 4, Life-threatening consequences: urgent intervention indicated. Grade 5, Death related to AE.
To evaluate changes in vital signs in healthy male participants, following a single oral dose of LIB-01. | 14 days
  Clinically significant changes in vital signs (blood pressure, pulse, respiratory rate, body temperature).
To evaluate changes in ECG in healthy male participants, following a single oral dose of LIB-01. | 14 days
  Clinically significant changes in ECG parameters (resting heart rate [HR] and PQ/PR, QRS, QT and QTcF intervals).
To evaluate the incidence of treatment-emergent adverse events as assessed by CTCAE in healthy male participants, following multiple oral dosing of LIB-01. | 28 days
  Frequency, seriousness and intensity of adverse events. Adverse events will be graded from 1-5 by the Common Terminology Criteria for Adverse Events (CTCAE):
  Grade 1, Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2, Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL).
  Grade 3, Severe or medically significant but not immediately life-threatening; hospitalisation or prolongation of hospitalisation indicated; disabling; limiting self- care ADL.
  Grade 4, Life-threatening consequences: urgent intervention indicated. Grade 5, Death related to AE. Clinically significant changes in vital signs, ECG and safety laboratory measurements.
To evaluate changes in vital signs in healthy male participants, following a multiple oral dosing of LIB-01. | 28 days
  Clinically significant changes in vital signs (blood pressure, pulse, respiratory rate, body temperature).
To evaluate changes in ECG in healthy male participants, following multiple oral dosing of LIB-01. | 28 days
  Clinically significant changes in ECG parameters (resting heart rate [HR] and PQ/PR, QRS, QT and QTcF intervals).

SECONDARY OUTCOMES:
To characterise the maximum plasma concentration of LIB-01, following a single oral dose. | 3 days
  Maximum Plasma Concentration [Cmax]
To characterise the plasma concentration half life of LIB-01, following a single oral dose. | 3 days
  Plasma Concentration Half Life [T1/2]
To characterise the plasma concentration area under curve of LIB-01, following a single oral dose. | 3 days
  Plasma Concentration Area Under Curve [AUC]
To characterise the maximum plasma concentration of LIB-01 following multiple oral dosing. | 4 days
  Maximum Plasma Concentration [Cmax]
To characterise the plasma concentration half life of LIB-01 following multiple oral dosing. | 4 days
  Plasma Concentration Half Life [T1/2]
To characterise the plasma concentration half life of LIB-01 following multiple oral dosing. | 4 days
  Plasma Concentration Area Under Curve [AUC]

CONTACTS AND LOCATIONS:
Overall Officials: Björn Schultze, MD, Principal Investigator — CTC
Locations (1):
- Clinical Trial Consultants, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No